CLINICAL TRIAL: NCT04487574
Title: A Multicenter, Adaptive, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of XC221, Tablets, 100 mg in Patients With COVID-19
Brief Title: A Study to Assess the Efficacy and Safety of XC221 in Patients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RSV Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XC221-03-02-2020
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: SARS-CoV-2 Infection
Keywords: COVID19; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — XC221

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Tablets identical in terms of composition, appearance and labeling to XC221 tablets, but without active substance will be used as Placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XC221 (Experimental): XC221 100 mg orally.
  1 tablet of XC221 100 mg 2 times a day during 14 days of treatment period.
  Interventions: Drug: XC221
- Placebo (Placebo Comparator): Placebo orally.
  1 tablet of Placebo 2 times a day during 14 days of treatment period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XC221 — Participants will receive XC221 100 mg 2 times a day during 14 days
  Arms: XC221
Drug: Placebo — Participants will receive Placebo 2 times a day during 14 days
  Arms: Placebo

SUMMARY:
The innovative drug XC221 100 mg tablet is designed for the treatment of COVID-19 (SARS-CoV-2 infection). A multicenter, adaptive, randomized, double-blind, placebo-controlled Phase III clinical study is aimed to assess the efficacy and safety of XC221 100 mg tablet, in COVID-19 patients during a 14-day treatment.

The primary objective of the study is to demonstrate the efficacy of XC221 100 mg tablet (200 mg daily dose) in achieving clinical improvement of COVID-19 symptoms.

The secondary objective of the study is to evaluate the safety of XC221 100 mg tablet (200 mg daily dose) in COVID-19 patients.

DETAILED DESCRIPTION:
11 Russian centers will participate in this study. The trail will consist of three periods: screening (duration not more than 1 day, it may coincide with the randomization visit and beginning of drug administration), treatment period (14 days) and follow-up period (14 ± 1 days after completion of treatment with XC221 / Placebo). The duration of participation in the study for each patient will be no more than 30 days.

118 eligible patients with confirmed COVID-19 will be randomized into two groups (Group A and Group B) in a 1:1 ratio: Group A - XC221 200 mg daily (59 patients); Group В - Placebo (59 patients).

During the treatment period (14 days), 1 tablet of XC221 / Placebo will be administered 2 times a day in addition to the standard of care (SoC) for COVID-19 according to The Temporary guidelines for the prevention, diagnosis and treatment of SARS-CoV-2 infection of the Ministry of Health of the Russian Federation (the MoH Temporary Guidelines). The follow-up period will last for 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form.
2. Patients of both sexes aged 18 to 75 years inclusive.
3. Diagnosed COVID-19 based on:

   * positive laboratory tests confirming the SARS-CoV-2 presence, performed no earlier than 14 days before hospitalization. It is allowed to determine the SARS-CoV-2 by the PCR or by another method according to the MoH Temporary Guidelines; and / or
   * bilateral alterations in lungs, typical for COVID-19, according to CT scan of the chest.
4. Patients with moderate or severe form of disease (t > 38.0°C; respiratory rate (RR) >22 / min; Sp02 <95%) not requiring non-invasive / invasive ventilation and / or high-flow oxygenation (HFNT), and / or extracorporeal membrane oxygenation (EMO) at the time of screening and randomization (based on the MoH Temporary Guidelines).
5. Patients requiring oxygen therapy (oxygenation through a nasal cannula, a simple facemask or other similar oxygen delivery device) with a category "4" according to the WHO scale.
6. Time from hospitalization to the first drug administration should not exceed 48 hours. This item is to be assessed only when re-evaluating the inclusion / exclusion criteria at the Randomization visit and treatment initiation.
7. Disease duration is no more than 7 full days since the moment of appearing one or more of the symptoms below until the first dose of the drug administration:

   * temperature increase;
   * dry cough or cough with little phlegm;
   * shortness of breath;
   * myalgia;
   * fatigue;
   * feeling of congestion in the chest;
   * reduced sense of smell and / or taste.
8. For women only: negative pregnancy test result. Pregnancy testing is not required for women of not childbearing potential (WONCBP): women who are in menopause (defined as an absence of menstruation for at least 2 years or more), or women who undergone surgical sterilization (hysterectomy, bilateral oophorectomy, tubal ligation), or women with a clinical diagnosis of "infertility". The presence of surgical sterilization and infertility should be confirmed by patient's claim or by relevant document confirming this condition.
9. Consent to use reliable method of contraception throughout the study period.
10. Patients who are able to understand and comply with treatment and procedures during the study.

Exclusion Criteria:

1. Known or suspected hypersensitivity to the active substance or to excipients of the drug XC221 or placebo
2. Known or suspected hypersensitivity to standard therapy drugs specified in The MoH Temporary Guidelines.
3. Lactase deficiency, lactose intolerance, glucose-galactose malabsorption.
4. Presence or suspicion of oncological diseases by the day of criteria assessment or in medical history (within the last 2 years).
5. Presence of autoimmune diseases by the day of criteria assessment or in medical history.
6. Neutropenia (0.5 * 10^9 /l).
7. Exceeding the upper limit of normal for ALT and AST by 5 times or more.
8. Thrombocytopenia 50000 / mm^3.
9. Pregnancy.
10. Lactation.
11. Presence of serious lung diseases, including, but not limited to the following diseases: moderate and severe bronchial asthma, severe and extremely severe COPD, interstitial lung disease, pulmonary hypertension, pulmonary fibrosis, surgical interventions on the lungs, tuberculosis (including suspicion of tuberculosis based on the results of CT examination at screening).
12. Patients with type 1 diabetes mellitus and / or decompensated type 2 diabetes mellitus.
13. Heart failure, NYHA functional class III - IV.
14. Chronic liver failure stage II (decompensated) and higher.
15. The need of renal replacement therapy at the time of inclusion of the patient.
16. Organ transplantation in medical history.
17. Medical history of epilepsy or the need for anticonvulsant therapy.
18. Major depressive disorder, anxiety, other mental disorders requiring medical correction.
19. Acute cerebrovascular accident, stroke or transient ischemic attack within 90 days before screening.
20. Administration of any antiviral and / or immunomodulatory drugs after the manifestation of COVID-19, with the exception of those specified in the MoH Temporary Guidelines.
21. Any immunosuppressive therapy (including tocilizumab / sarilumab) within 90 days prior to randomization, or the need of immunosuppressive therapy at the time of randomization.
22. Administration of systemic glucocorticosteroids within 90 days prior to randomization, or the need of systemic glucocorticosteroids at the time of randomization.
23. Administration of vaccines against viral infections within 90 days prior to randomization.
24. Patients receiving other experimental drugs, drugs not approved in the Russian Federation, or participating in other clinical trials within 30 days before screening.
25. Patients abusing alcohol or psychotropic drugs and other drugs by the day of criteria assessment or during the last year.
26. Patients with other serious, unstable, or clinically significant medical or psychological conditions that, in the opinion of the investigator, may preclude the patient's participation in the study.
27. Expected death within 48 hours after randomization.
28. Expected hospital discharge within 48 hours of randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-07-25 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Patient rate with a transition to category 3 or lower according to the WHO scale by Day 14 after the beginning of drug administration. | Day 1 - Day 14
  The scale of the patient's clinical condition, proposed by the WHO, will be used to assess the severity of patient general condition. Ranges for patient's clinical condition: 0 points (no infection) - 8 points (death).

SECONDARY OUTCOMES:
Time till clinical improvement, which is described by presence of all of the following factors during 48 hours in a row. | Day 1 - Day 28
  * Body temperature ≤ 37.5°C without using NSAIDs and / or paracetamol;
  * RR ≤ 22 / min without oxygen therapy;
  * SpO2 ≥ 95% without oxygen therapy.
Patient rate with clinical improvement by day 2-28. Presence of all of the following factors during 48 hours in a row. | Day 1 - Day 28
  * Body temperature ≤ 37.5°C without using NSAIDs and / or paracetamol;
  * RR ≤ 22 / min without oxygen therapy;
  * SpO2 ≥ 95% without oxygen therapy.
Patient rate with a negative test result for SARS-CoV-2 by Day 7±1, 15±1, 21 ±1 and 28 ± 1. | Day 1 - Day 28
Duration of hospitalization. | Day 1 - Day 28
Patient rate transferred to the intensive care unit (ICU) during hospitalization. | Day 1 - Day 28
Duration of ICU stay. | Day 1 - Day 28
Patient rate with ARDS during hospitalization. | Day 1 - Day 28
Presence of a fatal outcome. | Day 1 - Day 28
Patient rate requiring oxygen therapy by Day 2-28. | Day 1 - Day 28
Patient rate requiring high-flow oxygen therapy by Day 2-28. | Day 1 - Day 28
Patient rate requiring non-invasive ventilation by Day 2-28. | Day 1 - Day 28
Patient rate requiring invasive ventilation by Day 2-28. | Day 1 - Day 28
Patient rate requiring extracorporeal membrane oxygenation (EMO) by Day 2-28. | Day 1 - Day 28
The total duration of oxygen therapy by the last day of hospitalization. | Day 1 - Day 28
The total duration of high-flow oxygen therapy by the last day of hospitalization. | Day 1 - Day 28
The total duration of non-invasive ventilation by the last day of hospitalization. | Day 1 - Day 28
The total duration of invasive ventilation of lungs by the last day of hospitalization. | Day 1 - Day 28
The total duration of EMO by the last day of hospitalization. | Day 1 - Day 28
Patient rate with Sp02 > 95% by Day 2-28. | Day 1 - Day 28
Average alteration of Sp02 by Day 2-28 from baseline. | Day 1 - Day 28
Average time to reach SpO2 ≥ 95%. | Day 1 - Day 28
Patient rate with RR < 22 / min by Day 2-28. | Day 1 - Day 28
Average alteration in RR by Day 2-28 from baseline. | Day 1 - Day 28
Average time to reach RR ≤ 22 / min. | Day 1 - Day 28
Patient rate with body temperature < 37.5°C by Day 2-28. | Day 1 - Day 28
Average alteration in body temperature by Day 2-28 from baseline. | Day 1 - Day 28
Average time until the patient reaches a body temperature of ≤37.5°C. | Day 1 - Day 28
Patient rate with CT-1 according to CT data by Day 2-28. | Day 1 - Day 28
Average alteration in CT data by 1 point in terms of severity (CT-1, CT-2, CT-3, CT-4) by Day 7, 10, 15, 18, 21 and 28 compared to the baseline value. | Day 1 - Day 28
Average time to reach CT-1 according to CT data. | Day 1 - Day 28
Patient rate with a score < 2 according to the Daytime and Nighttime Cough Scale by Day 2-28. | Day 1 - Day 28
  The Daytime and Nighttime Cough Scale will be used to assess the dynamics of cough during the study. Ranges for assess: 0 points (no cough) - 6 points (severe cough that makes daytime activity impossible).
Mean change in Daytime and Nighttime Cough scores by Day 2-28 from baseline. | Day 1 - Day 28
  The Daytime and Nighttime Cough Scale will be used to assess the dynamics of cough during the study. Ranges for assess: 0 points (no cough) - 6 points (severe cough that makes daytime activity impossible).
Average time to reach < 2 points when assessed according to the Daytime and Nighttime Cough Scale. | Day 1 - Day 28
  The Daytime and Nighttime Cough Scale will be used to assess the dynamics of cough during the study. Ranges for assess: 0 points (no cough) - 6 points (severe cough that makes daytime activity impossible).
Patient rate with a score < 1 for each symptom (general fatigue, chest congestion, sore throat, decreased sense of smell and taste, nasal congestion) according to a 4-point scale by Day 2-28. | Day 1 - Day 28
  The Symptom Rating Scale will be used to assess the individuals' subjective ratings the severity of 6 symptoms of COVID-19. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 18 points) is a sum of points for each symptom.
Average change in score for each symptom (general fatigue, chest congestion, sore throat, decreased sense of smell and taste, nasal congestion) according to a 4-point scale by Day 2-28 from baseline. | Day 1 - Day 28
  The Symptom Rating Scale will be used to assess the individuals' subjective ratings the severity of 6 symptoms of COVID-19. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 18 points) is a sum of points for each symptom.
Average time to reach a score of < 1 for each symptom (general fatigue, feeling of congestion in the chest, sore throat, decreased sense of smell and taste, nasal congestion) according to a 4-point scale. | Day 1 - Day 28
  The Symptom Rating Scale will be used to assess the individuals' subjective ratings the severity of 6 symptoms of COVID-19. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 18 points) is a sum of points for each symptom.
Patient rate with a transition decrease to category 3 or lower according to the WHO scale by Day 2-13 and Day 15-28. | Day 1 - Day 28
  The scale of the patient's clinical condition, proposed by the WHO, will be used to assess the severity of patient general condition. Ranges for patient's clinical condition: 0 points (no infection) - 8 points (death).
Mean WHO grade change by Day 2-28 from baseline. | Day 1 - Day 28
  The scale of the patient's clinical condition, proposed by the WHO, will be used to assess the severity of patient general condition. Ranges for patient's clinical condition: 0 points (no infection) - 8 points (death).
Average time to reach the 3rd category or below according to the WHO scale. | Day 1 - Day 28
  The scale of the patient's clinical condition, proposed by the WHO, will be used to assess the severity of patient general condition. Ranges for patient's clinical condition: 0 points (no infection) - 8 points (death).
Patient rate with a NEWS score < 2 by Day 2-28. | Day 1 - Day 28
  Parameters will be assessed according to the National Early Warning Score only during hospitalization. During the treatment period, the assessment will be performed 2 times a day. During the follow-up period, the assessment will be performed once a day. The worst result for each period is to be chosen.
Average change in NEWS score by Day 2-28 from baseline. | Day 1 - Day 28
  Parameters will be assessed according to the National Early Warning Score only during hospitalization. During the treatment period, the assessment will be performed 2 times a day. During the follow-up period, the assessment will be performed once a day. The worst result for each period is to be chosen.
Average time to reach a NEWS score ≤ 2. | Day 1 - Day 28
  Parameters will be assessed according to the National Early Warning Score only during hospitalization. During the treatment period, the assessment will be performed 2 times a day. During the follow-up period, the assessment will be performed once a day. The worst result for each period is to be chosen.

OTHER OUTCOMES:
Concentration of IL-6 on Days 3 ± 1, 7 ± 1, 15 ± 1. | Day 1 - Day 15
  (Search Outcome)

CONTACTS AND LOCATIONS:
Locations (5):
- Russia (5):
  - Municipal Budgetary Institution of Healthcare "Central City Hospital of Novoshakhtinsk", Novoshakhtinsk, Rostov Oblast
  - Saint Petersburg State Budgetary Institution of Healthcare "City Hospital No. 40 of Kurortny District", Saint Petersburg
  - Saint Petersburg State Budgetary Institution of Healthcare "City Pokrovskaya Hospital" (4th Cardiology Department), Saint Petersburg
  - Saint Petersburg State Budgetary Institution of Healthcare "City Pokrovskaya Hospital", Saint Petersburg
  - Regional State Budgetary Institution of Healthcare "Medical-Sanitary Unit No. 2", Tomsk

IPD SHARING:
Plan to Share IPD: No